CLINICAL TRIAL: NCT05768958
Title: Hedonic and Homeostatic Appetite Control in Obesity and Type 2 Diabetes in the Context of Meal and Exercise Timing
Acronym: TIMEX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University of Leeds (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-22019913
Record Dates: First submitted 2023-02-15; First posted 2023-03-15 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Overweight and Obesity; Type 2 Diabetes
Keywords: Overweight; Obesity; Timing; Acute exercise; Circadian rythm; Appetite; Type 2 diabetes; Metabolism
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Morning exercise (Experimental): Study visit performed in the morning with 45 min exercise.
  Interventions: Other: Exercise
- Morning control (Experimental): Study visit performed in the morning with 45 min rest period.
  Interventions: Other: Control
- Evening exercise (Experimental): Study visit performed in the evening with 45 min exercise.
  Interventions: Other: Exercise
- Evening control (Experimental): Study visit performed in the evening with 45 min rest period.
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise — 45 min exercise bout performed on bicycle ergometer. The exercise bout will consist of a 10 min warm-up period at 40 % Watt max followed by 4 cycles of 4 min at 85 % Watt max and 3 min at 50 % Watt max. A cool-down period (7 min) will be performed at 40 % Watt max.
  Arms: Evening exercise; Morning exercise
Other: Control — 45 min rest during the same time period as the exercise bout on exercise study visits.
  Arms: Evening control; Morning control

SUMMARY:
The overall aim is to investigate effects of acute exercise on ad libitum energy intake and study whether this differs between morning and evening in individuals with overweight/obesity with or without type 2 diabetes (T2D). Furthermore, the aim is to examine the role of hedonic and homeostatic drivers of appetite control in obesity and T2D in the context of meal and exercise timing.

DETAILED DESCRIPTION:
Fifty-eight adults (age 18 - 75 years old) with overweight/obesity (BMI >25 kg/m2) and with/without T2D will participate in this randomized cross-over study. Participants will complete two visits in the morning and two in the evening with a minimum of 3 days washout. The visits will include ratings of subjective appetite and blood samples in the fasted state followed by either a 45 min exercise bout or rest for the same duration. 15 min after the termination of the exercise bout/rest period the participants will be presented with an ad libitum meal for assessment of energy intake (primary outcome). Then the participants will complete the Steno Biometric Food Preference Task (SBFPT); A computerized task measuring food choice, explicit liking, and implicit and explicit wanting with concomitant biometric measurements. Throughout the visits, subjective appetite will be rated using visual analogue scales and blood will be collected for assessment of appetite-related hormones and metabolites.

(Time: -60 minutes (fasting), -45 minutes (start exercise/rest), 0 minutes (finish exercise/rest), 15 minutes (ad libitum meal), 30 minutes (finish al libitum meal), 60 minutes (end of visit)

Descriptive data will be collected at a visit prior to the test days. These data include body weight (kg), Body Mass Index (BMI, kg/m2), fat mass (kg), fat free mass (kg), fat percentage (%), HbA1c (mmol/mol and %), waist circumference (cm), VO2-0peak and ECG. The participants will furthermore fill in questionnaires regarding the following: Socio-Economic Status (SES), Control Over Eating (CoEQ), Munich Chronotype Questionnaire (MCTQ), Physical Activity Questionnaires (IPAQ), Pittsburgh Sleep Quality Index (PSQI). In addition to the outcomes listed below, markers of liver function (Alanine aminotransferase (ALAT), Aspartate Transaminase (ASAT)), HbA1c, sodium, and potassium will be measured in the fasting state on the first morning visit.

The specific objectives are to:

1. Assess whether energy intake during an ad libitum meal differs after an acute bout of exercise compared to a rest condition
2. Assess whether energy intake during an ad libitum meal after an acute bout of exercise differs between morning and evening
3. Assess whether appetite ratings, food reward, and metabolic markers i.e., hormones and metabolites in response to an acute exercise bout and subsequent ad libitum meal differ between morning and evening
4. Examine if the above findings differ between individuals with and without T2D
5. Identify circulating biomarkers that can be used to stratify individuals with overweight/obesity into primary hedonic or homeostatic driven in terms of ad libitum food intake

ELIGIBILITY:
Inclusion Criteria:

* Adults with overweight or obesity (BMI >25 kg/m2) with and without T2D
* HbA1c ≥48 mmol/mol for people with T2D

Exclusion Criteria:

* Not able to eat ad libitum meal
* Not able to perform the exercise bout
* Daily smoking
* For women: Pregnancy / planned pregnancy (within the study period) / lactating
* Self-reported history of an eating disorder in the past 3 years
* Self-reported weight change (>5 kg) within three months prior to inclusion
* Treatment with antidepressants
* Treatment with fast acting insulin, combination insulin products and sulfonylureas
* Alcohol/drug abuse or in treatment with disulfiram (antabus) at time of inclusion
* Uncontrolled medical issues including but not limited to cardiovascular pulmonary, rheumatologic, hematologic, oncologic, infectious, gastrointestinal, or psychiatric disease; diabetes or other endocrine disease; immunosuppression
* Current treatment with medication which significantly affect appetite or energy balance (e.g., GLP-1 receptor agonists)
* Bariatric surgery
* Unable to understand the informed consent and the study procedures
* Concomitant participation in intervention studies
* Incapable of understanding Danish

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Ad libitum energy intake (KJ) after exercise compared with rest | Measured after meal consumption at t = 30 minutes
  Food intake (KJ) is measured after meal completion, exercise compared with rest

SECONDARY OUTCOMES:
Ad libitum energy intake (KJ) after exercise in the morning compared with evening | Measured after meal consumption at t = 30 minutes
  Assess whether energy intake during an ad libitum meal after exercise differs between morning and evening
Ad libitum energy intake (KJ) after rest in the morning compared with evening | Measured after meal consumption at t = 30 minutes
  Assess whether energy intake during an ad libitum meal after rest differs between morning and evening
Eating pace (KJ/min) | Measured from start to finish of meal consumption at t = 15 minutes to end of meal, morning and evening, exercise and rest
  Energy intake relative to duration of meal consumption
Glucose (mmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of glucose
Triglyceride (mmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of triglyceride
Total cholesterol (mmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of total cholesterol
LDL cholesterol (mmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of LDL cholesterol
HDL cholesterol (mmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of HDL cholesterol
VLDL cholesterol (mmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of VLDL cholesterol
Free-Fatty Acids (mmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of Free-Fatty Acids.
Circulating metabolides (metabolomics) (g/mL) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of circulating metabolides measured with metabolomic analysis
Circulating lipids (lipidomics) (g/mL) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of circulating lipids measured with lipidomic analysis
Circulating proteins (proteomics) (g/mL) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of circulating proteins measured with proteomic analysis
Insulin (pmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of insulin
Glucagon (pmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of glucagon
Total ghrelin (pmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of total ghrelin
Acylated ghrelin (pmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of acylated ghrelin
Glucagon-Like Peptide-1 (GLP-1) (pmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of Glucagon-Like Peptide-1 (GLP-1)
Glucose-Dependent Insulinotropic polypeptide (GIP) (pmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of Glucose-Dependent Insulinotropic polypeptide (GIP)
C-peptide (pmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of C-peptide
Peptide YY (PYY) (pmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of Peptide YY (PYY)
Peptide YY (PYY) 3-36 (pmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of Peptide YY (PYY) 3-36
Fibroblast Growth Factor 21 (FGF-21) (pmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of Fibroblast Growth Factor 21 (FGF-21)
Leptin (pmol/L) | Fasting (t = -60 minutes), and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of Leptin
Growth Differentiation Factor 15 (GDF-15) (pmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of Growth Differentiation Factor 15 (GDF-15)
Cholecystokinin (CCK) (pmol/L) | Fasting (t = -60 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of Cholecystokinin (CCK)
Pancreatic polypeptide (PP) (pmol/L) | Fasting (t = -60 minutes), and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of Pancreatic polypeptide (PP)
C-reactive protein (CRP) (pmol(L) | Fasting (t = -60 minutes), and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Concentrations of C-reactive protein (CRP)
Food choice | Measured before exercise/rest (t = -60 minutes) and after meal consumption (t= 30 minutes), morning and evening, exercise and rest
  Food choice of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the SBFPT. Food choice is determined based on frequency of selection made within each food category. The scores range from 0-48 i.e. 0 = foods within a specific food category have not been selected at all to 48 = foods within a specific food category have been selected 48 times.
Attention | Measured before exercise/rest (t = -60 minutes) and after meal consumption (t= 30 minutes), morning and evening, exercise and rest
  Measured using eye tracking in response to looking at food pictures during the computerized Leeds Food Preference Questionnaire.
  Includes the following parameters: Gaze: Time spent (ms and %) and revisits (n); and fixations: Time to first fixation (ms), time spent (ms and %), fixation count (n), first fixation duration (ms), average fixation duration (ms). Distance to screen (mm), and gaze direction bias (ratio) which is calculated as the number of trials in which the first fixation was directed to a food image as a proportion to all trials. A bias score ˃0.5 indicates attention towards one food image, a bias score equal to 0.5 indicates no bias, and a bias score <0.5 indicates attention towards the other food images.
Reaction time (ms) | Measured before exercise/rest (t = -60 minutes) and after meal consumption (t= 30 minutes), morning and evening, exercise and rest
  Reaction time during forced food choice of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the computerized Leeds Food Preference Questionnaire.
Explicit liking | Measured before exercise/rest (t = -60 minutes) and after meal consumption (t= 30 minutes), morning and evening, exercise and rest
  Explicit liking of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the SBFPT. Explicit liking is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how pleasant would it be to taste this food right now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Implicit wanting | Measured before exercise/rest (t = -60 minutes) and after meal consumption (t= 30 minutes), morning and evening, exercise and rest
  Implicit wanting of food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the SBFPT. Implicit wanting is assessed based on food choice and response time for selected and non-selected food items as well as mean response time (a frequency-weighted algorithm).
  In this frequency-weighted algorithm a positive score indicates a more rapid preference for a food type over another food type and a negative score indicates the opposite. A score of zero indicates that food types are equally preferred. The frequency weighted algorithm is used so the implicit wanting score is influenced by both selection (positively contributing to the score) and non-selection (negatively contributing to the score) of food type. Scores for implicit wanting typically range from -100-100 (due to reaction time there is no fixed min-max value)
Explicit wanting | Measured before exercise/rest (t = -60 minutes) and after meal consumption (t= 30 minutes), morning and evening, exercise and rest
  Explicit wanting of 16 food items from four combined food categories (high-fat savoury, high-fat sweet, low-fat savoury and low-fat sweet foods) examined from the SBFPT. Explicit wanting is rated using visual analogue scales and the range is 0-100. Each end represents the extremes e.g. Question: "how much do you want some of this food now?" Answer: "not at all" (rated 0 on the 0-100 scale) to "extremely" (rated 100 on the 0-100 scale).
Subjective appetite | Fasting (t = -60, 0 minutes) and at t = 0, 15, 30, 45, 60 minutes, morning and evening, exercise and rest
  Rated using visual analogue scales and includes sensations of: Hunger, fullness, satiety, prospective food consumption, wellbeing, nausea, thirst, desire to eat meat, salty, and sweet. The scale range is 0-100 and each end represent the extremes e.g. hunger rating: "I am not hungry at all" to "I have never been this hungry before".
Energy intake (KJ) | Registered 24 hours after the test days, morning and evening, exercise and rest
  Assessed from diet records
Borg RPE | Measured after exercise (t = 0 minutes) , morning and evening
  Subjective rating of the level of exertion during exercise is collected through the Borg Rating of Percieved Exertion (RPE) at baseline and post exercise, and compared between visits.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Færch, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data from the trial will not be made publicly available as individual data from participants are protected by EU's GDPR (General Data Protection Regulation) laws and Danish Data Protection laws. Study results can be made available upon reasonable request from the corresponding author.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Jalking L, Launbo NP, Jensen MM, Pedersen HE, Blond MB, Gerstenberg MK, Finlayson G, Beaulieu K, Faerch K, Grunnet LG, Quist JS. Effects of exercise and exercise timing on energy intake and appetite control in Danish individuals with overweight or obesity with and without type 2 diabetes: a protocol for a randomised controlled cross-over trial. BMJ Open. 2025 Feb 6;15(2):e092683. doi: 10.1136/bmjopen-2024-092683. PMID 39915022